CLINICAL TRIAL: NCT06890507
Title: The Anti-Anginal Effects of N-Acetylcysteine (NAC) in Patients with Angina and Non-Obstructive Coronary Arteries (ANOCA)
Acronym: NANA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Adelaide (Other)
Responsible Party: Principal Investigator, Sivabaskari Pasupathy, Post doctoral Research Fellow, University of Adelaide
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025/HRE00080
Record Dates: First submitted 2025-03-16; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Angina Attacks; Non Obstructive Coronary Artery Disease
Keywords: ANOCA; Angina with Non Obstructive Coronary Arteries; N-acetylcysteine
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Randomised, double-blind, placebo-controlled crossover study assessing the anti-anginal effect and impact on health status of NAC 600mg twice daily in patients with ANOCA experiencing angina at least 3 times/week32
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral NAC 600mg (twice daily) Intervention Arm (Experimental): This arm will assess the effects of oral N-Acetylcysteine (NAC) at a dose of 600mg twice daily in patients with ANOCA. Participants will receive the NAC treatment for a 4-week period.
  Interventions: Drug: N-Acetylcysteine (NAC)
- Placebo 600mg twice daily (Placebo Comparator): This arm will serve as the placebo comparator in the crossover study design. Participants will receive a placebo treatment that is identical in appearance to the NAC medication but contains no active ingredient.The order of treatment (NAC vs placebo) is randomized and participants remain blinded throughout the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-Acetylcysteine (NAC) — The investigational product for this study is NAC 600 mg capsules. The NAC drug substance is sourced from a Good Manufacturing Practice (GMP)-certified supplier by Syntro Health Pty Ltd and tested on receipt
  Arms: Oral NAC 600mg (twice daily) Intervention Arm
Drug: Placebo — To ensure appropriate blinding and to match the physical characteristics of the NAC capsules, the placebo capsules will be filled with dicalcium phosphate (DCP). DCP has been selected over microcrystalline cellulose due to the weight requirements of the NAC formulation.
  Arms: Placebo 600mg twice daily

SUMMARY:
The goal of this clinical trial is to determine if N-acetylcysteine (NAC) can reduce angina frequency in women with Angina with Non-Obstructive Coronary Arteries (ANOCA). It will also assess the impact of NAC on health status and quality of life. The main questions it aims to answer are:

(i) Does NAC reduce the number of angina episodes per week? (ii) How does NAC affect quality of life and symptom burden in ANOCA patients? (iii) Does NAC reduce the need for short-acting nitrate use?

Researchers will compare NAC to a placebo in a randomized, double-blind, placebo-controlled crossover study to determine its effectiveness.

Participants will receive treatment with NAC 600mg twice daily for 4 weeks (28 days) and matched placebo for 4 weeks (28 days) in a computer-generated random order giving a total dosing period of 8 weeks. There will be a 2-week washout between the two treatment periods.

The effectiveness of N-Acetylcysteine (NAC) will be assessed using the following measures:

Angina Diary: Participants will record the frequency and severity of their angina episodes.

Seattle Angina Questionnaire-7 (SAQ-7): Participants will complete this questionnaire to assess physical limitations, angina frequency, and quality of life.

EuroQol 5-Dimension (EQ-5D) Questionnaire: Participants will rate their overall health and quality of life.

DETAILED DESCRIPTION:
Background:

Angina with Non-Obstructive Coronary Arteries (ANOCA) refers to a condition where patients experience chronic angina despite having no significant coronary artery blockages. This condition affects 50-70% of women undergoing elective angiography, in stark contrast to just 7-17% of men. Many experience a prolonged delay in diagnosis, resulting in notable decreases in functional capacity.

NAC has been shown to reduce oxidative stress and potentiate the vasodilatory and antiaggregatory effects of nitrates, potentially reducing microvascular damage and improving myocardial perfusion, hence presenting a promising therapeutic option for ANOCA patients. Although there are no established clinical guidelines for ANOCA management, standard therapy typically includes both long-acting and short-acting nitrates to alleviate anginal symptoms. However, many ANOCA patients continue to experience symptoms despite standard therapy. As such, this trial will assess the beneficial effects of NAC therapy in ANOCA women.

Primary Objectives: To determine the effect of NAC 600mg twice daily on angina frequency in patients with ANOCA who experience angina at least 3 times/week as assessed by an angina diary.

Secondary Objective: The secondary objectives of this study are:

i. To assess the impact of NAC therapy (600mg twice daily) on quality of life/health status, utilising generic (EQ-5D) and disease-specific (SAQ-7) health status instruments to evaluate the following PROMs:

1. Overall physical health (EQ-5D)
2. Angina frequency (SAQ-7)
3. angina-related physical limitations (SAQ-7)
4. angina-related quality of life (SAQ-7)
5. patient satisfaction with angina therapy (SAQ-7) ii. To assess the impact of NAC therapy (600mg twice daily) on angina diary measures including:

a) Short-acting nitrate consumption (i.e., Glyceryl trinitrate (GTN) spray use) b) Duration of angina episodes c) Severity of angina episodes

Safety objectives i. Emergency Department (ED) presentations with Chest pain ii. Hospital admissions with chest pain iii. Major Adverse Coronary Events (MACE) Clinic Assessments: Visit 1: Screening: Screening assessments will be completed within 14 days prior to administration of NAC/Placebo.

* Consent to participate
* Baseline safety bloods (complete blood examination, electrolytes, liver & kidney functions tests, high sensitivity C-reactive protein, ionised calcium)
* Physical Examination
* Vital assessments
* Electrocardiogram (ECG) assessment Week 1 & 2
* Angina Diary Visit 2: Weeks 3-6: Phase 1 study medication period
* Angina Diary
* Health-related questionnaires (SAQ-7, EQ-5D) Visit 3: End of Phase 1 visit
* Angina Diary
* Health-related questionnaires (SAQ-7, EQ-5D) Weeks 7& 8 Wash out Period
* Angina Diary Visit 4: Weeks 9-12 Phase 2 study medication period
* Angina Diary
* Health-related questionnaires (SAQ-7, EQ-5D) Visit 5: End of Phase 2 visit
* Health-related questionnaires (SAQ-7, EQ-5D) Weeks 4,10 & 14 Follow up Phone Contact Duration of Therapy: Patients will receive treatment with NAC 600mg twice daily for 4 weeks (28 days) and matched placebo for 4 weeks (28 days) in a computer-generated random order (double-blind, crossover design) giving a total dosing period of 8 weeks. There will be a 2-week (14 day) washout between the two treatment periods.

Criteria for Evaluation: Angina diary: Results will be considered significant if participants have significantly (p<0.05) reduced features of angina extracted from angina diary during the NAC phase compared to placebo phase.

SAQ-7: Results will be considered significant if participants demonstrate reduced physical limitations & angina frequency and improved quality of life during NAC phase compared to placebo phase.

EQ-5D: Results will be considered significant if participants demonstrate improved quality of life scores during NAC Phase compared to placebo phase.

Statistical Methods: Efficacy Endpoint NAC's anti-anginal efficacy will be undertaken by blinded analysis of the angina diary endpoints and other endpoints. The comparison between patients with respect to treatment order will be analysed utilising a linear mixed-effects model.

Safety Endpoint Frequency and severity of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Female patients aged ≥18 years
3. No obstructive CAD (defined as either absence of epicardial lesions with ≥50% luminal narrowing in any coronary artery segment on coronary angiography or normal findings on computed tomography (CT) angiogram, indicating the absence of significant stenosis) to account for chest pain symptoms.
4. Chest pain occurring ≥3 times/week in the preceding two weeks.

Exclusion Criteria:

1. Known allergy to NAC or its components.
2. Acute myocardial infarction admission within the preceding month (hospital admission for prolonged angina paint associated with a cardiac troponin level above the 99th percentile, with a subsequent rise or fall).
3. Secondary causes of angina including:

i. clinically significant anaemia (haemoglobin <100g/dL) ii. uncontrolled atrial fibrillation (ventricular response rate >108bpm) iii. haemodynamically significant aortic stenosis (mean valve gradient ≥40mmHg) d) Known concomitant disease with life expectance of less than 1 year. e) Abnormalities in liver function tests suggesting hepatic impairment (ALT and/or AST 2 x upper limit of normal (ULN) or ALP 2 x ULN or Bilirubin 1.5 x ULN) f) Severe renal impairment (eGFR <30mL/min) or on dialysis. g) Pregnancy or lactation. h) Untreated hypertension i) Unwilling, or unable, to give informed consent, including due to severe psychiatric conditions affecting informed consent process or compliance.

j) History of substance abuse. k) Currently taking Chloroquine. l) Serious or unstable medical conditions that may interfere with the study, as determined by the PI.

m) Concomitant participation in another clinical trial or research study (except where in the opinion of the PI, the participant could benefit from enrolling in another trial)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female sex
Enrollment: 25 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of angina episodes recorded in angina diary. | 8 weeks (4 weeks of NAC treatment and 4 weeks of placebo treatment)
  Number of angina episodes recorded in angina diary. The angina diary is developed to record the frequency, duration, severity, and reliever of chest pain episodes. Participant record their angina episodes throughout the study period.

SECONDARY OUTCOMES:
Frequency of Short-acting nitrate consumption (i.e., Glyceryl trinitrate (GTN) spray use) | 8 weeks (4 weeks treatment compared to 4 weeks placebo)
  Short-acting nitrate consumption (i.e., Glyceryl trinitrate (GTN) spray use), self reported on angina diary
Frequency of prolonged angina episodes (ie episodes persisting > 20 minutes) | 8 weeks (4 weeks of NAC treatment and 4 weeks of placebo treatment)
  Frequency of prolonged angina episodes (ie episodes persisting > 20 minutes) assessed from patient's self reported angina diary
Angina frequency score as assessed by Seattle Angina Questionnaire (SAQ) | End of Phase 1 (Score at the end of 4 weeks) & End of Phase 2 ( Score at the end of 4 weeks)
  The Seattle Angina Questionnaire (SAQ) is a tool used to assess the health-related quality of life in patients with angina, especially those with coronary artery disease (CAD).
  Patients report the frequency of their angina episodes, including both exertional and spontaneous chest pain, based on structured response options. The score is then converted to a 0-100 scale, with higher scores indicating less frequent angina and better symptom control.
Angina-related physical limitations score as assessed on Seattle Angina Questionnaire | End of Phase 1 (Score at the end of 4 weeks) & End of Phase 2 ( Score at the end of 4 weeks)
  The Angina-Related Physical Limitations Score is a subscale of the Seattle Angina Questionnaire (SAQ) that evaluates the extent to which angina symptoms restrict a patient's ability to perform daily physical activities.
  Patients rate the difficulty they experience in performing activities such as walking, climbing stairs, or carrying groceries due to their angina. Responses are scored on a 0-100 scale, where higher scores indicate fewer physical limitations and better functional status.
Angina-related quality of life score as assessed on Seattle Angina Questionnaire | End of Phase 1 (Score at the end of 4 weeks) & End of Phase 2 ( Score at the end of 4 weeks)
  Patients assess the impact of angina on their overall quality of life, including emotional well-being, physical limitations, and social functioning. The score is converted to a 0-100 scale, with higher scores reflecting better quality of life and less impact from angina.
Patient satisfaction with angina therapy score as assessed on Seattle Angina Questionnaire | End of Phase 1 (Score at the end of 4 weeks) & End of Phase 2 ( Score at the end of 4 weeks)
  Patients rate their satisfaction with the current treatment regimen for managing angina, based on structured questions related to the effectiveness, convenience, and side effects of therapy. The score is converted to a 0-100 scale, with higher scores indicating greater satisfaction.
Overall physical health as assessed by EQ-5D Questionnaire | End of Phase 1 (Score at the end of 4 weeks) & End of Phase 2 ( Score at the end of 4 weeks)
  EQ-5D is a standardized questionnaire developed by the EuroQol Group to measure health-related quality of life.
  Patients assess their overall physical health through the EQ-5D, which includes questions related to mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The score is then converted to a 0-100 scale, with higher scores indicating better overall physical health and less impact from the condition.
Severity score of angina episodes as assessed on angina diary | 8 weeks (4 weeks of NAC treatment and 4 weeks of placebo treatment)
  Angina severity score (scored as 1-10), 10 being most intense assessed from patient's self-reported angina diary

CONTACTS AND LOCATIONS:
Overall Officials: John Beltrame, PhD, Principal Investigator — University of Adelaide; Sivabaskari Pasupathy, PhD, Principal Investigator — University of Adelaide
Locations (1):
- The Queen Elizabeth Hospital, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No
The collected data contains confidential patient health information. De-identified data may be made available upon request, but it will not be publicly accessible due to the inclusion of confidential patient health information. Access will be granted in accordance with ethical guidelines and institutional policies, ensuring that all requests are reviewed and approved before data is shared